CLINICAL TRIAL: NCT00433459
Title: First International Inter-Group Study for Classical Hodgkin's Lymphoma in Children and Adolescents
Brief Title: Combination Chemotherapy in Treating Young Patients With Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Christine Mauz-Körholz (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); Euronet Worldwide (Other)
Responsible Party: Sponsor-Investigator, Christine Mauz-Körholz, Prof. Dr. med. Christine Mauz-Körholz, Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000531687; EURONET-PHL-C1; EU-20703; EUDRACT-2006-000995-33; CCLG-HD-2007-10
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: childhood lymphocyte depletion Hodgkin lymphoma; childhood mixed cellularity Hodgkin lymphoma; childhood nodular sclerosis Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Cyclophosphamide; Dacarbazine; Prednisolone; Prednisone; Procarbazine; Vincristine; Fluorodeoxyglucose F18; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPP (Active Comparator): procarbazine-containing consolidation chemotherapy arm
  Interventions: Drug: cyclophosphamide; Drug: prednisolone; Drug: prednisone; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: fludeoxyglucose F 18; Radiation: radiation therapy
- COPDAC (Experimental): procarbazine-free consolidation chemotherapy arm
  Interventions: Drug: cyclophosphamide; Drug: dacarbazine; Drug: prednisolone; Drug: prednisone; Drug: vincristine sulfate; Radiation: fludeoxyglucose F 18; Radiation: radiation therapy

INTERVENTIONS:
Drug: cyclophosphamide — drug is used in first line treatment in combination (COPP or COPDAC)
  Other Names: CYC
Drug: dacarbazine — drug is used in first line treatment in combination (COPDAC)
  Other Names: DTIC
  Arms: COPDAC
Drug: prednisolone — drug is used in first line treatment in combination (OEPA, COPP or COPDAC)
Drug: prednisone — drug is used in first line treatment in combination (OEPA, COPP or COPDAC)
Drug: procarbazine hydrochloride — drug is used in first line treatment in combination (COPP)
  Arms: COPP
Drug: vincristine sulfate — drug is used in first line treatment in combination (OEPA, COPP or COPDAC)
  Other Names: VCR
Radiation: fludeoxyglucose F 18 — used as a diagnostic marker for metabolically active tumour at staging and response assessment
Radiation: radiation therapy — part of combination treatment (combined modality between chemo- and radiotherapy)
  Other Names: IFRT

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective in treating Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying different combination chemotherapy regimens to compare how well they work in treating young patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the 5-year event-free survival (EFS) rate in pediatric patients with Hodgkin's lymphoma with an adequate response after 2 courses of vincristine, etoposide, prednisone, and doxorubicin hydrochloride (OEPA) (without radiotherapy) are consistent with an estimated target EFS rate of 90%.
* Compare the EFS (without a deterioration) of patients treated with procarbazine hydrochloride vs dacarbazine (treatment groups 2 and 3).
* Determine the treatment outcome of a standardized risk-adapted relapse strategy in these patients.

Secondary

* Determine whether the 5-year EFS rate in patients with Hodgkin's lymphoma with an inadequate response after 2 OEPA courses and standard involved-field radiotherapy are consistent with an estimated target EFS rate of 90%.
* Determine whether a positive positron emission tomography scan before planned high-dose chemotherapy with autologous stem cell transplantation has a negative prognostic significance.
* Compare the effect of dacarbazine vs procarbazine on the rate of infertility in males and premature menopause in females (treatment groups 2 and 3).

Tertiary

* Determine the impact of real-time central staging and response assessment on treatment outcome in these patients.

OUTLINE: This is a randomized, controlled, parallel-group, open-label, multicenter study. Patients are stratified according to staging and response assessment (central vs local) and disease stage (IA/B or IIA [first-line treatment group 1] vs I_EA/B, II_EA, IIB, or IIIA [first-line treatment group 2] vs II_EB, III_E A/B, IIIB, or IVA/B [first-line treatment group 3]).

* First-line treatment group 1: Patients receive oral prednisone (or prednisolone) 3 times daily on days 1-15, vincristine IV on days 1, 8, and 15, doxorubicin hydrochloride IV over 1-6 hours on days 1 and 15, and etoposide (or etoposide phosphate) IV over 1-2 hours on days 1-5 (OEPA).

Treatment repeats every 28 days for 2 courses in the absence of unacceptable toxicity. Patients are assessed by fludeoxyglucose F 18 positron emission tomography (^18FDG-PET) scan. Patients with inadequate response undergo radiotherapy within 35 days after completion of OEPA.

* First-line treatment group 2: Patients receive OEPA as in group 1. After completion of OEPA, patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral prednisone (or prednisolone) 3 times daily and oral procarbazine hydrochloride 2-3 times a day on days 1-15 and vincristine IV and cyclophosphamide IV over 1 hour on days 1 and 8 (COPP).
  * Arm II: Patients receive oral prednisone (or prednisolone) 3 times daily on days 1-15, dacarbazine IV over 15-30 minutes on days 1-3, and vincristine IV and cyclophosphamide IV over 1 hour on days 1 and 8 (COPDAC).

In both arms, treatment repeats every 28 days for 2 courses in the absence of unacceptable toxicity. Patients are assessed by ^18FDG-PET scan. Patients with an inadequate response undergo radiotherapy within 35 days after completion of COPP or COPDAC.

* First-line treatment group 3: Patients receive OEPA as in group 1. After completion of OEPA, patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive COPP as in arm I of group 2.
  * Arm II: Patients receive COPDAC as in arm II of group 2. In both arms, treatment repeats every 28 days for 4 courses in the absence of unacceptable toxicity. Patients are assessed by ^18FDG-PET scan. Patients with an inadequate response undergo radiotherapy within 35 days after completion of COPP or COPDAC.

Patients with biopsy-confirmed disease progression OR relapse after first-line treatment on this study or on protocols DAL-HD 90, GPOH-HD 95, GPOHHD 2002 Pilot, or similar treatment proceed to second-line therapy. Patients are stratified according to relapse/progression status (late relapse from first-line treatment group 1 [second-line treatment group 1] vs early relapse from first-line treatment groups 1, 2, or 3 or late relapse from first-line treatment groups 2 or 3 [second-line treatment group 2] vs disease progression [second-line treatment group 3]). Patients undergo a ^18FDG-PET scan prior to beginning second-line therapy.

* Second-line treatment group 1: Patients receive ifosfamide IV over 22 hours and etoposide IV over 1-2 hours and oral prednisone three times daily on days 1-5 (IEP). Patients then receive doxorubicin hydrochloride IV over 1-6 hours, bleomycin IV, vinblastine IV, and dacarbazine IV over 15-30 minutes on days 22 and 36 (ABVD). Treatment repeats every 50 days for 2 courses in the absence of disease progression or unacceptable toxicity.

After chemotherapy treatment, patients undergo radiotherapy.

* Second-line treatment group 2: Patients receive IEP and ABVD as in group 1. Autologous stem cells are collected after course 1 or 2 of IEP/ABVD.

After chemotherapy, patients with an adequate response undergo radiotherapy. Patients with an inadequate response undergo high-dose chemotherapy comprising carmustine IV over 1-2 hours on day -7, etoposide IV and cytarabine IV over 30 minutes twice daily on days -6 to -3, and melphalan IV over 1½ hours on day -2. Patients then undergo autologous hematopoietic stem cell transplantation (HSCT).

Patients undergo a ^18FDG-PET scan on day 50-54. Patients with ^18FDG-PET scan positive disease undergo radiotherapy.

* Second-line treatment group 3: Patients receive IEP and ABVD as in group 1. All patients then undergo high-dose chemotherapy and HSCT as in group 2.

Patients undergo a ^18FDG-PET scan on day 50-54. Patients with ^18FDG-PET scan positive disease undergo radiotherapy.

After completion of study therapy, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 2,150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classical Hodgkin's lymphoma

  * No lymphocyte-predominant Hodgkin's lymphoma
  * Fine-needle biopsy not sufficient
* No prior treatment for Hodgkin's lymphoma except for recommended pre-phase therapy for a large mediastinal tumor

PATIENT CHARACTERISTICS:

* No known hypersensitivity or contraindication to study drugs
* No other current malignancy
* No severe concurrent disease (e.g., immune deficiency syndrome)
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for up to 1 year after completion of study treatment
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy
* At least 30 days since prior and no other concurrent investigational drugs or participation in another investigational trial

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2134 (Actual)
Dates: Start 2007-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Progression-free survival | 5 years
CTC (Common toxicity criteria) toxicity levels of therapy elements | 5 years
Evidence of male infertility score | 5 years
Evidence of female infertility score | 5 years
Long-term consequences (e.g., premature menopause, secondary cancer) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Koerholz, MD, Study Chair — Martin-Luther-Universität Halle-Wittenberg; W. Hamish Wallace, MD, Principal Investigator — Royal Hospital for Sick Children; Judith Landman-Parker, MD, Principal Investigator — Hopital d'Enfants Trousseau
Locations (2):
- Universitaetsklinikum Giessen-Marburg, Giessen, Germany
- Royal Hospital for Sick Children, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Daw S, Claviez A, Kurch L, Stoevesandt D, Attarbaschi A, Balwierz W, Beishuizen A, Cepelova M, Ceppi F, Fernandez-Teijeiro A, Fossa A, Georgi TW, Hjalgrim LL, Hraskova A, Leblanc T, Mascarin M, Pears J, Landman-Parker J, Prelog T, Klapper W, Ramsay A, Kluge R, Dieckmann K, Pelz T, Vordermark D, Korholz D, Hasenclever D, Mauz-Korholz C. Transplant and Nontransplant Salvage Therapy in Pediatric Relapsed or Refractory Hodgkin Lymphoma: The EuroNet-PHL-R1 Phase 3 Nonrandomized Clinical Trial. JAMA Oncol. 2025 Mar 1;11(3):258-267. doi: 10.1001/jamaoncol.2024.5636. PMID 39745682
- [Derived] Pabari R, McCarten K, Flerlage J, Lai H, Mauz-Korholz C, Dieckmann K, Palese M, Kaste S, Castellino SM, Kelly KM, Stoevesandt D, Kurch L. Hodgkin lymphoma involving the extra-axial CNS: an AHOD1331, PHL-C1, and PHL-C2 report from the COG and EuroNet-PHL. Blood Adv. 2024 Sep 24;8(18):4856-4865. doi: 10.1182/bloodadvances.2023012346. PMID 39058968
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- [Derived] Mauz-Korholz C, Landman-Parker J, Fernandez-Teijeiro A, Attarbaschi A, Balwierz W, Bartelt JM, Beishuizen A, Boudjemaa S, Cepelova M, Ceppi F, Claviez A, Daw S, Dieckmann K, Fossa A, Gattenlohner S, Georgi T, Hjalgrim LL, Hraskova A, Karlen J, Kurch L, Leblanc T, Mann G, Montravers F, Pears J, Pelz T, Rajic V, Ramsay AD, Stoevesandt D, Uyttebroeck A, Vordermark D, Korholz D, Hasenclever D, Wallace WH, Kluge R. Response-adapted omission of radiotherapy in children and adolescents with early-stage classical Hodgkin lymphoma and an adequate response to vincristine, etoposide, prednisone, and doxorubicin (EuroNet-PHL-C1): a titration study. Lancet Oncol. 2023 Mar;24(3):252-261. doi: 10.1016/S1470-2045(23)00019-0. PMID 36858722
- [Derived] Mauz-Korholz C, Landman-Parker J, Balwierz W, Ammann RA, Anderson RA, Attarbaschi A, Bartelt JM, Beishuizen A, Boudjemaa S, Cepelova M, Claviez A, Daw S, Dieckmann K, Fernandez-Teijeiro A, Fossa A, Gattenlohner S, Georgi T, Hjalgrim LL, Hraskova A, Karlen J, Kluge R, Kurch L, Leblanc T, Mann G, Montravers F, Pears J, Pelz T, Rajic V, Ramsay AD, Stoevesandt D, Uyttebroeck A, Vordermark D, Korholz D, Hasenclever D, Wallace WH. Response-adapted omission of radiotherapy and comparison of consolidation chemotherapy in children and adolescents with intermediate-stage and advanced-stage classical Hodgkin lymphoma (EuroNet-PHL-C1): a titration study with an open-label, embedded, multinational, non-inferiority, randomised controlled trial. Lancet Oncol. 2022 Jan;23(1):125-137. doi: 10.1016/S1470-2045(21)00470-8. Epub 2021 Dec 9. PMID 34895479
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/about-cancer/treatment/clinical-trials/search/v?a=8&id=NCI-2014-02026&loc=0&rl=2&st=C7258&t=C9357